CLINICAL TRIAL: NCT01181414
Title: Phase 4. Study of Cardiac Resynchronization Therapy in Patients With Permanent Atrial Fibrillation.
Brief Title: Spanish Atrial Fibrillation And Resynchronization Study
Acronym: SPAREIII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Navarrra Hospital (Clinica Universitaria) (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario La Fe (Other); Hospital Universitario La Paz (Other); Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of the Arrhythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPARE III - 2010
Record Dates: First submitted 2010-08-02; First posted 2010-08-13 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Heart Failure; Cardiomyopathy, Dilated; Atrial Fibrillation
Keywords: Permanent Atrial Fibrillation; Resynchronization therapy; Ablation
MeSH Terms: conditions — Cardiomyopathy, Dilated; Atrial Fibrillation | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrioventricular junction ablation (Experimental): Atrioventricular junction ablation by using radiofrequency energy.
  Interventions: Procedure: Atrio ventricular junction ablation with radio-frequency
- Drug control of ventricular rate (Active Comparator): Drug control of ventricular rate.
  Interventions: Drug: Beta blocker/digoxine/amiodarone

INTERVENTIONS:
Procedure: Atrio ventricular junction ablation with radio-frequency — Atrioventricular junction ablation by using radiofrequency energy.
  Arms: Atrioventricular junction ablation
Drug: Beta blocker/digoxine/amiodarone — Ventricular rate control by using drug treatment.
  Other Names: Negative chronotropic drugs pharmacological treatment .
  Arms: Drug control of ventricular rate

SUMMARY:
The aim of the present study is to compare the response to cardiac resynchronization therapy (CRT) in patients with chronic advanced heart failure and permanent atrial fibrillation (AF) depending on atrio ventricular junction (AVJ) is ablated or not.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) improves the functional capacity and the quality of life and reduces the mortality of patients with dilated cardiomyopathy, low ejection fraction and wide QRS.

Only 2% of patients included in CRT randomized trials were in AF.

To obtain a good response to CRT, percentage >90% of ventricular pacing must be obtained.

Based on observational studies, current guidelines of CRT recommend the atrio ventricular junction (AVJ) ablation in those patients with permanent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy (LVEDD >56 mm)
* wide QRS (> 120 msec)
* NYHA III-IV
* EF<35%
* Permanent AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular reverse remodelling in cardiac resynchronization therapy and atrial fibrillation. | 1-year follow-up
  Comparison of echocardiographic responders in patients with permanent atrial fibrillation submitted to cardiac resynchronization therapy depending on whether the atrio-ventricular junction is ablated or not. Echocardiographic response was defined as left ventricular end-systolic volume reduction >10%.

SECONDARY OUTCOMES:
Clinical response to Cardiac resynchronization therapy. | 1-year follow-up
  Comparison of clinical response in patients with permanent atrial fibrillation submitted to cardiac resynchronization therapy, depending on whether the atrio-ventricular junction has been ablated or not. Clinical response is defined as not death/heart transplantation and improvement of the distance walked in the 6-minute walking test >10%.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Tolosana, M.D., Principal Investigator — Hospital Clinic, University of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain